CLINICAL TRIAL: NCT04237038
Title: Long-term Quality of Life Results After Laparoscopic Fundoplication With and Without Short Gastric Vessel Division in Gastroesophageal Reflux Management
Brief Title: Quality of Life Results After Laparoscopic Fundoplication.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Clinical Professor, Instituto Mexicano del Seguro Social
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R-2013-601-8
Record Dates: First submitted 2019-11-28; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Quality of Life
Keywords: Laparoscopic fundoplication; Short gastric vessel

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial was conducted with patients submitted to laparoscopic Nissen fundoplication between February 2013 to december 2014 according to the guidelines established by the Mexican Consensus for the study of GERD.
Masking Description: Assignment to the treatment or control group was provided with random numbers in sealed envelopes conducted by a physician of the outpatient clinic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- laparoscopic Nissen fundoplication short gastric vessel divi (Experimental): Randomized clinical trial conducted in forty patients submitted to short gastric vessel division (SGVD) forty patients without SGVD. Patients were evaluated with standarized questionnaires to measure the degree of satisfaction in relation to surgical procedure and to the quality of life.
  Interventions: Procedure: laparoscopic Nissen fundoplication short gastric vessel division

INTERVENTIONS:
Procedure: laparoscopic Nissen fundoplication short gastric vessel division — Randomized clinical trial conducted in forty patients submitted to SGVD and forty patients without SGVD. Patients were evaluated with standarized questionnaires to measure the degree of satisfaction in relation to surgical procedure and to the quality of life. A randomized clinical trial was conducted with 87 patients submitted to laparoscopic Nissen fundoplication between February 2013 to december 2014 according to the guidelines established by the Mexican Consensus for the study of Gastroesophageal reflux disease (GERD

SUMMARY:
The present study focuses on determining aspects of satisfaction and quality of life of patients that underwent laparoscopic Nissen fundoplication with or without short gastric vessel division (SGVD) and long-term differences.

DETAILED DESCRIPTION:
The aim of our study was to identify the degree of satisfaction and the quality of life of patients that underwent laparoscopic Nissen total fundoplication with or without SGVD.

Materials and methods. A randomized clinical trial was conducted with 87 patients submitted to laparoscopic Nissen fundoplication between February 2013 to december 2014 according to the guidelines established by the Mexican Consensus for the study of GERD.12 Inclusion criteria: 1) Patients who underwent surgery against Gastroesophageal Reflux with Nissen Fundoplication by Laparoscopic Pathway who were not divided into short gastric vessels during the procedure. 2) Patients who underwent surgery against Gastroesophageal Reflux with Nissen Fundoplication by Laparoscopic Route who underwent a division of short gastric vessels during the procedure. 3) Operated between October 2003 and November 2011 at the General Hospital of Zone # 1 "Dr. Leonel Ramírez García "of the IMSS Colima delegation. Exclusion criteria: 1)Patients in whom conversion to open surgery was performed. 2) Operated before October 2003 or after November 2011.3) Patients whose data is not available for their location. Disposal criteria:1) Patients not reachable for any reason.2. Patients who do not wish to participate. 3. Patients with incomplete medical information for research.

The patients were assigned into two groups: 43 patients that had SGVD and 44 patients in whom the short gastric vessels were left intact. Seven patients were lost during the follow-up, leaving 40 patients in the SGVD group and 40 in the group without SGVD. The mean follow-up time was 5±0,5 years (4 to 6 years) and the Nissen total fundoplication was the only surgical procedure performed by the authors. Complications, hospital stay, and surgical time (secondary aims) were identified in a blinded fashion. The time it took to return to daily activities, the degree of satisfaction measured, quality of life, and symptom persistence (primary aims) were identified through standardized questionnaires that were previously validated for that purpose. The level of satisfaction, quality of life of the postopera-tive patients, and surgical morbidity were evaluated through standardized and validated questionnaires elaborated for that purpose. The Carlsson questionnaire was applied to all the patients in order to measure reflux intensity; quality of life was studied postoperatively through the GIQLI (an adequate,valid,and useful instrument for evaluating quality of life in patients presenting with reflux disease)because it includes specific questions about digestive symp-toms and generic questions about physical,emotional,and social capacity.The questionnaire contains 36 items with an answer scale from0(the worst result) to 4(the best result).Global scores above 86 were regarded as a satisfactory effect, even in the presence of residual symptoms.Dysphagia was evaluated with the Dysphagia score,the Analog scale for dysphagia,and the Visick grading system.The questionnaire dealing with the level of satisfaction and quality of life was applied to each patient that had a minimum5-year postoperative period; it was applied verbally and the questions were asked by a researcher uninvolved in the surgical management.The level of satisfaction was evaluated nominally with the following questions:Would you accept being operated on again? Would you recommend the procedure to a friend or familymember? TheGIQLI was chosen because it is a validated questionnaire n Spanish.It consists of 36 questions divided in to 5 sections,with a specific part for digestive diseases.Scoring and the visual analog for dysphagia were measured through validated sco-ring scales,whereas the Visick scale was measured ordinally.

Statistical analysis. A database was designed (Microsoft Excel) and the statistical analysis was done through the IBM SPSS Statistics ver. 21 (©copyright IBM Corporation) program. The comparative analysis of the groups was carried out under the principles of intention-to-treat. Descriptive statistics were used as mean, standard deviation and percentages. The comparison of averages between groups was performed using Student t or Mann-Whitney U tests (for equal variances or different respectively). The percentage comparison was made with Chi-square or Fisher exact tests. While the pairwise comparison of ordinal variables Wilcoxon test was used. In all statistical test, a confidence interval of 95% was used. Statistical significance was set at a p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients who underwent surgery against Gastroesophageal Reflux with Nissen Fundoplication by Laparoscopic Pathway who were not divided into short gastric vessels during the procedure.
* 2) Patients who underwent surgery against Gastroesophageal Reflux with Nissen Fundoplication by Laparoscopic Route who underwent a division of short gastric vessels during the procedure.
* 3) Operated between October 2003 and November 2011 at the General Hospital of Zone # 1 "Dr. Leonel Ramírez García "of the IMSS Colima delegation.

Exclusion Criteria:

* 1) Patients who underwent surgery against Gastroesophageal Reflux with Nissen Fundoplication by Laparoscopic Pathway who were not divided into short gastric vessels during the procedure.
* 2) Patients who underwent surgery against Gastroesophageal Reflux with Nissen Fundoplication by Laparoscopic Route who underwent a division of short gastric vessels during the procedure.
* 3) Operated between October 2003 and November 2011 at the General Hospital of Zone # 1 "Dr. Leonel Ramírez García "of the IMSS Colima delegation.

Ages: 22 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Carlsson questionnaire | five years
  Carlsson questionnaire was applied to all the patients in order to measure reflux intensity. A total score between -7 and +18 points is obtained. Consider a score greater than or equal to 4 as positive for GERD.
Gastrointestinal Quality of Life Index (GIQLI) Gastrointestinal Quality of Life Index: GIQLI Gastrointestinal Quality of Life Index: GIQLI | five years
  evaluating quality of life in patients presenting with reflux disease.The maximum GIQLI in the international score is 144 and its worst value is 0
Visick grading system | five years
  Scale used to assess the assessment of patients regarding antireflux surgery, both openly and laparoscopically. The patient globally assesses the subjective outcome of the surgery: 1 = cured / asymptomatic, 2 = improved / scarce symptoms without the need for medical treatment, 3 = no significant changes / symptoms that require medical treatment, and 4 = worsened / great symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIO PRIETO DIAZ-CHAVEZ, PhD, Study Director — Universidad de Colima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Prieto-Diaz-Chavez E, Medina-Chavez JL, Brizuela-Araujo CA, Gonzalez-Jimenez MA, Mellin-Landa TE, Gomez-Garcia TS, Gutierrez-Zamora J, Trujillo-Hernandez B, Millan-Guerrero R, Vasquez C. Patient satisfaction and quality of life following laparoscopic Nissen fundoplication. Rev Gastroenterol Mex. 2014 Apr-Jun;79(2):73-8. doi: 10.1016/j.rgmx.2013.11.003. Epub 2014 May 27. English, Spanish. PMID 24878219
- See also: http://dx.doi.org/10.1016/j.rgmx.2013.11.003 — http://dx.doi.org/10.1016/j.rgmx.2013.11.003